CLINICAL TRIAL: NCT05215743
Title: Cardioprotection of Patients With Acute Myocardial Infarction Undergoing Percutaneous Coronary Angioplasty Through a Combined Antioxidant Therapy. A Phase I, Randomized Clinical Trial.
Brief Title: Combined Antioxidant Therapy Against Myocardial Reperfusion Injury. Phase I Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, Ramon Rodrigo, Full Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FONDECYT 1211850
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Acute Myocardial Infarction; Ischemia-reperfusion Injury; Reperfusion Injury, Myocardial; Reperfusion Arrhythmias; Reperfusion Injury
Keywords: antioxidants; acute myocardial infarction; reperfusion injury; randomized clinical trial; multi-target interventions
MeSH Terms: conditions — Reperfusion Injury; Myocardial Reperfusion Injury | interventions — Acetylcysteine; Deferoxamine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Combined antioxidant therapy (CAT) and placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined antioxidant therapy (CAT) (Experimental): Intravenous administration of deferoxamine, n-acetylcysteine, and ascorbate over 90 minutes.
  Interventions: Drug: Antioxidant therapy
- Placebo (Placebo Comparator): Intravenous administration of NaCl 0.9% over 90 minutes
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Antioxidant therapy — Active therapy
  Other Names: ascorbate; n-acetylcysteine; deferoxamine
  Arms: Combined antioxidant therapy (CAT)
Drug: NaCl 0.9% — Placebo
  Other Names: saline solution
  Arms: Placebo

SUMMARY:
Background: Acute myocardial infarction (AMI) has remained a leading cause of mortality and disability worldwide. Although percutaneous coronary angioplasty (PCA) is the best treatment for these patients, paradoxically this procedure causes reperfusion injury. Considerable efforts aimed to reduce this damage have been made, but the results are disappointing and there is still no effective therapy for preventing the damage. Previously, the investigators have achieved a reduction of infarct size in an experimental model of an isolated rat heart, through a synergistic effect of three compounds in a "combined antioxidant therapy" (CAT).

In this study, the investigators aim to describe the pharmacokinetics and safety of CAT intravenously administered to healthy subjects. This is the first step to a later clinical application of CAT in AMI patients.

Methodology: The safety and pharmacokinetics of the CAT (deferoxamine, N-acetylcysteine, and ascorbate) will be assessed in healthy volunteers in a "phase I clinical trial". Two different formulations (mass of CAT components by bag) with different infusion rates each one will be tested (CAT1 and CAT2). Subjects (18-35 years old, n=18) will be randomized 1:2 to receive a placebo or CAT for 90 minutes. Blood concentrations of each CAT component will be measured in plasma at 0, 15, 30, 60, 90, 120, and 180 minutes after the infusion onset. Adverse events will be registered from the onset of infusion until day 30.

DETAILED DESCRIPTION:
In this single-blind trial, healthy subjects from 18-35 years old will be allocated to a placebo or an intravenous combined antioxidant therapy (CAT) following a fixed-dose scalation approach. Before the study onset, blood samples will be drawn from eligible subjects to measure a general health profile, and also a physician evaluation and medical exams will be scheduled to further confirm the healthy status two weeks after the CAT/placebo infusion.

Two different CAT formulations (named CAT1 and CAT2) will be tested, each one with a different dose of deferoxamine, N-acetylcysteine, and ascorbate. The infusions (CAT or placebo) will be administered at the "CREA" - Hospital Clínico Universidad de Chile. The first nine subjects will be randomized 1:2 to placebo (NaCl 0.9%) or CAT1, infused at two different rates (one in the first 30 min, and another one in the following 60 minutes). If the stopping rules are not observed (see below), then the next nine subjects will be randomized 1:2 to placebo or CAT2 to be infused I.V over 90 min at a constant rate. The protocol will be stopped at any time if more than 33% of the subjects in a group (2 volunteers) suffer a serious adverse event, following the international definitions (death, disability, life-threatening, medical admission).

Vital signs will be continuously assessed during the IV infusion and for the following 90 minutes after the infusion ends, together with adverse events assessment in this 180-minute observation period. Blood samples will be collected at 0, 15, 30, 60, 90, 120, and 180 minutes. Concentrations of ascorbate, deferoxamine, and N-acetylcysteine will be measured, as well as oxidative stress biomarkers. Subjects will be contacted by phone asking for health status and adverse events at 14 and 30 days after the IV infusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects from 18 to 35 years old
* Not obese (BMI 19-29.9 kg/m2)

Exclusion Criteria:

* Impaired renal function (creatinine > 1.5 mg/dL)
* Liver impairment (liver enzymes more than 3 times over normal values)
* Glucose 6-phosphate dehydrogenase deficiency
* Any chronic disease
* Any acute disease in the last two weeks
* To be enrolled in another clinical study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of each CAT component | 180 minutes (just before the infusion onset up to 90 minutes after infusion ending)
  Cmax of deferoxamine, n-acetylcysteine and ascorbate
Half-life time (T1/2) of each CAT component | 180 minutes (just before the infusion onset up to 90 minutes after infusion ending)
  T1/2 of deferoxamine, n-acetylcysteine and ascorbate
Area under the plasma concentration versus time curve (AUC) of each CAT component | 180 minutes (just before the infusion onset up to 90 minutes after infusion ending)
  AUC of deferoxamine, n-acetylcysteine and ascorbate
Volume of distribution (Vd) of each CAT component | 180 minutes (just before the infusion onset up to 90 minutes after infusion ending)
  Vd of deferoxamine, n-acetylcysteine and ascorbate
Clearence (CL) of each CAT component | 180 minutes (just before the infusion onset up to 90 minutes after infusion ending)
  CL of deferoxamine, n-acetylcysteine and ascorbate
Elimination rate constant (Ke) of each CAT component | 180 minutes (just before the infusion onset up to 90 minutes after infusion ending)
  Ke of deferoxamine, n-acetylcysteine and ascorbate
Incidence of serious adverse events during combined antioxidant therapy infusion or along the 30-day follow-up | From day 0 to day 30 after the intervention
  Number of new events that began during I.V infusion, the 90 minutes of observation after the infusion end, or during the 30-day follow-up, and that resulted in death, disability, life-threatening, or medical admission of a patient according to medical records

SECONDARY OUTCOMES:
Incidence of any adverse event (serious and non-serious) up to thirty days after infusion ending | From day 0 to day 30 after the intervention
  Number of serious and non-serious adverse events from day 0 to day 30 after the intervention, assessed by a phone interview on day 14 and day 30 after the infusion, using a standardized report form
Number of patients with any adverse event (severe and non-severe) up to thirty days after infusion ending | From day 0 to day 30 after the intervention
  Number of patients with serious and non-severe adverse events from day 0 to day 30 after the intervention, assessed by a phone interview on day 14 and day 30 after the infusion, using a standardized report form
Plasma levels of oxidative stress biomarkers over the time | 0 (just before infusion onset) and 30, 90 and120 minutes after infusion onset.
  Plasma concentrations of the antioxidant defenses (ferric reducing ability of plasma assay), and lipid peroxidation (F2-isoprostanes) during the IV infusion and after 30 minutes
Plasma concentrations over the time of each CAT component | 0 (just before infusion onset) and 30, 60, 90, 120 and 180 minutes after infusion onset.
  Plasma concentrations of deferoxamine, n-acetylcysteine and ascorbate during the IV infusion and after 90 minutes, assessed by high performance liquid chromatography (HPLC)

CONTACTS AND LOCATIONS:
Overall Officials: Ramón Rodrigo, Prof., Study Director — Program of Pharmacology, ICBM, Faculty of Medicine, University of Chile; Abraham IJ Gajardo, MD, PhD, Study Chair — Intensive Care Unit, Hospital Clínico Universidad de Chile
Locations (1):
- University of Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No